CLINICAL TRIAL: NCT05967767
Title: Three Sessions of Repeated Sprint Training in Normobaric Hypoxia With 48-Hour Interval Improves Repeated Sprint Performance Indices
Brief Title: Repeated Sprint Training in Normobaric Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Abdulkadir Birol, Assistant Professor, Trabzon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Interventional
Record Dates: First submitted 2023-07-15; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Hypoxia
Keywords: normobaric hypoxia; repeated sprint training
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: single-blind placebo-controlled design
Who Masked: Participant
Masking Description: In this study, blinding was provided in practice by using the simulation device for the normoxia condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3 Session Repeated Sprint Training in Normobaric Hypoxia (Experimental): Hypoxia group was exposed to normobaric hypoxia equal to 3420 m (FiO2: 13.5-13.6 %).
  Interventions: Device: Normobaric Hypoxia Exposure
- 3 Session Repeated Sprint Training in Normobaric Normoxia (Sham Comparator): Placebo group was exposed to normobaric normoxia equal to 162 m (FiO2: 20.9 %) through wearing the altitude generator mask.
  Interventions: Device: Normobaric Normoxia Exposure
- Control group (No Intervention): The control group was subjected to only pre and post-test.

INTERVENTIONS:
Device: Normobaric Hypoxia Exposure — Hypoxia group were exposed to normobaric hypoxia equal to 3420 m (FiO2: 13.5-13.6 %).
  Arms: 3 Session Repeated Sprint Training in Normobaric Hypoxia
Device: Normobaric Normoxia Exposure — Placebo group were exposed to normobaric normoxia equal to 162 m (FiO2: 20.9 %) through wearing the altitude generator mask.
  Arms: 3 Session Repeated Sprint Training in Normobaric Normoxia

SUMMARY:
The aim of the current study was to examine the effects of 3-session repeated sprint training performed in a normobaric hypoxic condition with 48-hour rest intervals on sprint performance indices, arterial oxygen saturation (SpO2) and rating of perceived exertion (RPE) scores. Twenty-four moderately-trained males participated in this study voluntarily basis. This study was conducted on single-blind placebo-controlled design. Participants were divided into three groups as follows; normobaric hypoxia (3420 m; HYP), normobaric normoxia (162 m; PLA) and control group (CON). HYP and PLA groups subjected to 3 repeated sprint training session (4 set x 5 x 5 s sprints with 30 s recovery and 5 min rest between the sets) in normobaric hypoxia or normoxia condition. Pre- and pos-test were conducted 72 hours before and after the training intervention period. All the training and testing sessions performed in cycle ergometer. There were no detected significant time and condition interaction in the variables; relative peak power output (PPO), mean power output (MPO), percentage of sprint decrement score (Sdec%) and RPE observed in the scope of pre- and post-test.

DETAILED DESCRIPTION:
This single-blind placebo-controlled designed study was approved by Ankara University Human Research Ethics Committee (2020/277) and conducted in accordance with the Declaration of Helsinki. The participants in normobaric hypoxia (HYP) and placebo (PLA) groups visited the laboratory six times and the control (CON) group visited three times. At the first visit of participants, the aim and the possible outcomes of the research was explained, the familiarization process for cycle ergometer and test/training protocol was performed, and the informed consent forms were obtained. The participants were divided randomly into three groups after the anthropometric measurements and baseline tests were completed so as part of the second visit. The groups were divided as follows; HYP group (n=9) which were exposed to normobaric hypoxia equal to 3420 m (FiO2: 13.5-13.6 %), PLA (n=7) that were exposed to normobaric normoxia equal to 162 m (FiO2: 20.9 %) through wearing the altitude generator mask, and the control group (CON; n=8) which was subjected to only pre and post-test. The determined hypoxic dose for HYP group was directly implemented (setting 9 was equal to 3420 m on used hypoxia generator), and no correction was made for the actual altitude (900 m, Golbasi, Ankara, Türkiye). The normobaric hypoxia and placebo condition was provided by Everest Summit II-Altitude Generator (Hypoxico Hypoxicator, New York, USA). At the 3rd-5th visits, HYP and PLA groups performed 3 repeated sprint training sessions under normobaric hypoxia or normoxia exposure with 48-hour intervals. And the participants visited the laboratory last time for post-test measurements. Each participant visited the laboratory for training sessions and test trials at the same time in the day. In the scope of pre and post-test repeated sprint indices, SpO2 and RPE data were collected. Pre-test and post-test were conducted 72 hours before and 72 hours after the training intervention period in normobaric normoxia condition. Including the testing days, the intervention period lasted 11 days in November 2022. All the experimental processes were conducted in Ankara University Performance Laboratory.

ELIGIBILITY:
Inclusion Criteria:

* non-smokers,
* male gender,
* those who do not have any chronic disease,
* do not use any medication,
* do not any training or accommodate above 1500 m altitude within the past 3 months,
* do not have any musculoskeletal injuries within the past 6 months and,
* train at least 3 days in a week.

Exclusion Criteria:

* Having a chronic or acute condition/disease during the intervention period
* Occurrence of acute respiratory illness or musculoskeletal injury during the intervention period
* Leaving the study voluntarily/on his own account

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Relative Peak Power Output | 11 days
  Relative peak power output (as newton meter) produced during the repeated cycling sprint tests by the participant in the scope of pre and post tests were recorded and assessed via Lode Cycling Ergometer Software. The total intervention period was 11 days from pre to post test. The change evaluated from pre to post test.
Relative Mean Power Output | 11 days
  Relative mean power output (as newton meter) produced during the repeated cycling sprint tests by the participant in the scope of pre and post tests were recorded and assessed via Lode Cycling Ergometer Software. The total intervention period was 11 days from pre to post test. The change evaluated from pre to post test.
Percentage of Sprint Decrement Score | 11 days
  Percentage of sprint decrement score calculated via relative peak power output produced during the repeated cycling sprint tests by the each participant in the scope of pre and post tests. The used sprint decrement score formula was as the follows; "Sdec% = [1 - (total power/ideal power)] × 100". Total power refers to accumulated PPO over the number of sprints and ideal power is defines the achieved highest PPO over the repetitions. An increase in the obtained score means that the sprint performance decreases.The total intervention period was 11 days from pre to post test. The change evaluated from pre to post test.

SECONDARY OUTCOMES:
Arterial Oxygen Saturation | 11 days
  Arterial oxygen saturation was measured and recorded via fingertip oximeter during the repeated cycling sprint tests for the end of the each sprint. The total intervention period was 11 days from pre to post test. The change evaluated from pre to post test.
Rate of Perceived Exertion | 11 days
  Rate of Perceived exertion evaluated via 6-20 Borg scale and recorded during the repeated cycling sprint tests for the end of the each sprint. The total intervention period was 11 days from pre to post test. The change evaluated from pre to post test.
  Scoring Level of Exertion 6 No Exertion 7 Extremely Light 8 9 Very Light 10 11 Light 12 13 Somewhat Hard 14 15 Hard (Heavy) 16 17 Very Hard 18 19 Extremely Hard 20 Maximal Exertion

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)